CLINICAL TRIAL: NCT00328380
Title: A Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety of Rifaximin for the Prevention of Travelers' Diarrhea in Subjects Traveling Outside the United States
Brief Title: Prevention of Travelers' Diarrhea in Subjects Traveling Outside the U.S.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RFID3004
Record Dates: First submitted 2006-05-17; First posted 2006-05-19 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Diarrhea
Keywords: Travelers' Diarrhea; Xifaxan; Rifaximin; Escherichia coli; E coli; EAEC; Enteroaggregative E coli; ETEC; Enterotoxigenic E coli
MeSH Terms: conditions — Diarrhea; Escherichia coli Infections | interventions — Rifaximin

INTERVENTIONS:
Drug: Rifaximin

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of rifaximin 600 mg (3 x 200-mg tablets) once daily compared with placebo when taken for 14 days by healthy subjects to prevent travelers' diarrhea (TD) from all causes.

DETAILED DESCRIPTION:
Travelers' diarrhea (TD) is the most common illness in travelers to the developing world, occurring in 60% or more of international travelers to high-risk areas. It can be quite debilitating for the usual 2 to 4 days of the illness and may lead to disruption of travel plans. Findings from recent studies have indicated that the chronic post-travel illness may prove to be of greater clinical and public health significance than the acute illness. Specifically, persistent diarrhea has been reported in 2% to 10% of travelers developing diarrhea. Moreover, bacterial enterocolitis, including that associated with TD, leads to post-infectious irritable bowel syndrome in 4% to 31% of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is in good health (as determined by medical history)
2. Subject is planning on traveling anywhere outside the US (except Canada) for at least 5 and no more than 14 days
3. Subject is scheduled to depart on their planned trip no later than 14 days and no earlier than 4 days after having blood drawn for clinical laboratory assessments and urine collected for a pregnancy test (females of childbearing potential only)

Exclusion Criteria:

1. Subject has hypersensitivity or allergy to rifaximin or rifampin
2. Subject has known or suspected alcohol abuse or illicit drug use within 1 year of enrollment
3. Subject participated in an investigational drug or device study within the 30 days prior to enrollment
4. Subject received rifaximin in a previous clinical study
5. Subject received any systemic or gastrointestinal-specific antibiotic within 7 days of the first dose of study drug
6. Subject received antidiarrheal medication (eg, loperamide, lactobacillus, BSS, Kaopectate®) within 24 hours of the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2005-12; Primary Completion 2006-12 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in this study is the assessment of safety and tolerability of rifaximin 600 mg QD compared to placebo.

SECONDARY OUTCOMES:
A secondary endpoints of this study include assessment of the differences between the 2 treatment groups based upon the proportion of subjects with TD during the 14-day Treatment Period.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Sunshine Medical Center, South Miami, Florida
  - Southwest Doctors, PA, Houston, Texas
  - La Porte Family Clinic, La Porte, Texas